CLINICAL TRIAL: NCT04977375
Title: Phase Ib/II Trial of Anti-PD-1 Immunotherapy and Stereotactic Radiation in Patients With Recurrent Glioblastoma
Brief Title: Trial of Anti-PD-1 Immunotherapy and Stereotactic Radiation in Patients With Recurrent Glioblastoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chirag G. Patil (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Chirag G. Patil, Associate Professor of Neurosurgery Program Director, Neurosurgery Residency Training, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2019-13-Patil-NeoPD1SRS; R21CA256421 (NIH)
Record Dates: First submitted 2021-04-22; First posted 2021-07-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma Multiforme
Keywords: Central Nervous System Tumor; neurosurgery; Brain tumor; spinal cord tumor; surgical resection; glioma; glioblastoma; neuropathology; maximal safe resection; CNS
MeSH Terms: conditions — Glioblastoma; Central Nervous System Neoplasms; Brain Neoplasms; Spinal Cord Neoplasms; Glioma | interventions — pembrolizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab with stereotactic radiation therapy and surgical resection (Experimental)
  Interventions: Drug: Pembrolizumab; Radiation: Stereotactic Radiation Therapy; Procedure: Surgical Resection

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 400mg administered intravenously on Day 1, and then beginning 6 weeks post-surgery, subjects will receive 400 mg pembrolizumab every 6 weeks
Radiation: Stereotactic Radiation Therapy — Standard of care stereotactic radiation of 24 grays over 3 days, administered beginning on Day 7
Procedure: Surgical Resection — Standard of care surgical resection of tumor on Day 10-28

SUMMARY:
The purpose of this study is to assess the safety/tolerability/feasibility of pembrolizumab and radiation therapy before surgical resection in patients with recurrent glioblastoma as defined by treatment-related AEs and the number of patients who do not necessitate a delay in surgical resection, and to assess overall survival. The secondary objectives are to assess progression free survival, and to assess the T cell clonality, CD8 T cell activation and Tumor Infiltrating Lymphocyte (TIL) score after treatment

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Confirmed histologic diagnosis of WHO Grade IV, Glioblastoma Multiforme
* GBM recurrence or progression with planned standard of care surgical resection and repeat radiation
* Tumor size less than 6 cm
* ECOG performance status of 0-1
* Adequate laboratory values

Exclusion Criteria:

* Contraindication to additional radiation
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor
* Immunodeficiency diagnosis or receiving chronic systemic steroid therapy (exceeding 10 mg daily of prednisone) or any other form of immunosuppressive therapy
* Severe hypersensitivity to pembrolizumab

Complete inclusion/exclusion criteria are detailed in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability measured by the incidence of adverse events, serious adverse events and grade 3 or above treatment related adverse events. | From start of study treatment until confirmation of disease progression, intolerable toxicities, withdrawal of consent. Assessed up to 2 years.
  Safety and tolerability measured by the incidence of adverse events, serious adverse events and grade 3 or above treatment related adverse events as assessed per CTCAE, Version 5.0.
Overall survival | From start of study treatment until death, loss to follow-up, or withdrawal of consent. Assessed up to 2 years.
  From start of study treatment until death, loss to follow-up, or withdrawal of consent. Subjects who are lost to survival follow-up will not be replaced, and public records may be accessed to assess Overall Survival.

SECONDARY OUTCOMES:
Progression free survival | From start of study treatment until until confirmation of disease progression, intolerable toxicities, withdrawal of consent. Assessed up to 2 years.
  From start of study treatment until confirmation of disease progression (per iRANO Criteria), intolerable toxicities, withdrawal of consent, or up to 2 years or 18 cycles of pembrolizumab, whichever comes first.
Immune action | At baseline, prior to stereotactic radiation therapy, and prior to surgery.
  To assess the T cell clonality, CD8 T cell activation and Tumor Infiltrating Lymphocyte (TIL) score after treatment. Blood draws for research purposes performed after obtaining consent but prior to neoadjuvant pembrolizumab administration, and at the time of initiation of SRT and at the time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chirag G Patil, MD, MS, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT04977375/ICF_000.pdf